CLINICAL TRIAL: NCT00892307
Title: Coronary Anatomy and Physiology Using Multidetector Dual Source Computed Tomography With Adenosine Enhancement: Comparative Study With SPECT Imaging: Pilot Studies I/II
Brief Title: Adenosine Dual Source Computed Tomography (CT) Versus Adenosine Single Photon Emission Computed Tomography (SPECT)
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel S. Berman, Principal Investigator, Cedars-Sinai Medical Center
Other Study IDs: IRB # 10928/11143
Record Dates: First submitted 2009-04-24; First posted 2009-05-04 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: Diagnostic Imaging; Dual Source Multidetector Computed Tomography; Computed Tomography; CT; Single Photon Emission Computed Tomography; SPECT; Myocardial Perfusion; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Dual Source Multidetector CT (DSCT) w/ Adenosine enhancement — Somatom Definition Dual Source CT Scanner Stress/Rest Image scan using weight based CT contrast dye
  Other Names: Dual Source Multidetector Computed Tomography; Dual Source CT; Dual Source CT with adenosine enhancement; Adenosine enhanced CT; Siemens Somatom Definition Dual Source Scanner

SUMMARY:
Researchers hope that this new non-invasive multi-detector scanner (DSCT) will provide diagnostic information comparable to the combination of traditional SPECT (for function and blood flow) and CT imaging (for a precise anatomical view).

DETAILED DESCRIPTION:
The DSCT scanner is able to assess cardiac blood flow (myocardial perfusion) at the same time as coronary anatomy. The results derived from these scans will be compared to standard SPECT imaging.

To further evaluate obstruction in the coronary arteries, physicians may refer for an invasive Coronary Angiogram, the current gold standard for diagnosis of Coronary Artery Disease (CAD). By validating the DSCT scanner as a system with which to assess the extent of obstruction in the coronary arteries, physicians may be able to lessen the occurrence of an invasive exam.

Procedures: Each pilot anticipates enrolling 20 subjects.

Pilot 1: Clinical Follow-up Rest/Stress Adeno-SPECT and Research Stress /Rest Adeno-DSCT obtained in the same patient during the same period of stress testing

* Radiation: Thallium injection for rest SPECT
* Drug: Single dose Adenosine Infusion for DSCT and SPECT
* Radiation: Sestamibi injection for stress SPECT
* Drug: CT contrast
* Radiation: Stress DSCT /Rest DSCT

Pilot 2: Research Stress/ Rest Adeno-DSCT obtained within 30 days of initial positive SPECT finding

* Drug: Adenosine Infusion for DSCT
* Drug: CT contrast
* Radiation: Stress DSCT /Rest DSCT

Both pilot studies will relate results to subject history, ECG and cardiac angiogram, if available

ELIGIBILITY:
Pilot 1:

Inclusion Criteria:

* Provide written consent and are willing to comply with protocol requirements
* Are at least 18 years of age
* Are referred for clinically-ordered SPECT
* Have known CAD

Exclusion Criteria:

* Patients being referred to invasive coronary angiography will not be included in this pilot
* Caffeine intake within the 24 hours prior to adenosine stress testing
* Pregnancy (known or suspected)
* Intolerance or contraindication to adenosine (severe Asthma…)
* Intake of methylxanthine containing medications such as theophylline that have not been withdrawn and would interfere with the effectiveness of adenosine.
* Unstable coronary syndromes
* Uncontrolled congestive cardiac failure or cardiogenic shock
* Uncontrolled hypertension with resting BP > 200/110
* More than 30 days between the Adeno-SPECT and the Adeno-DSCT
* Revascularization (percutaneous coronary intervention or coronary artery bypass graft surgery) between the Adeno-SPECT and the Adeno-DSCT
* Change in clinical status as determined by the investigator
* Inability to be on same medication regime 24 hrs prior to Adeno-SPECT and Adeno DSCT
* Patients with chronic renal failure (C.C.T. < 60 ml/m2/sec)
* Patients with allergy to contrast iodinated media
* Congestive heart failure
* History of thromboembolic disorders
* Multiple myeloma
* Hyperthyroidism
* Pheochromocytoma
* Atrial fibrillation
* Inability to perform breath hold for 12 seconds

Pilot 2:

All inclusions/exclusions are the same as Pilot 1, WITH THE ADDITION OF:

Inclusion Criteria:

* Have had prior (within 30 days) positive Adeno-SPECT scan

Exclusion Criteria:

* Patients with contraindications to coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary Artery Disease
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To show that adenosine enhanced DSCT will enhance regular Multidetector Spiral Computed Tomography (MSCT) "diagnostic power" to detect significant (e.g., > 50%) coronary stenosis | One day

SECONDARY OUTCOMES:
To assess coronary anatomical results obtained by CT Angiography (CTA) at high heart rates in terms of the rate of assessable coronary segments. | One day

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Berman, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States